CLINICAL TRIAL: NCT05619978
Title: A Multi-Center Retrospective Chart Review Study Examining the Patient Characteristics, Treatment Patterns, Clinical Outcomes, and Burden of Illness Among Patients With Chronic Myeloid Leukemia in Third-line Treatment or With T315I Mutation in France (CML 3L+ & T315I)
Brief Title: French Study to Highlight the Unmet Treatment Needs of 3L+ CP-CML and With T315I-mutated CML Patients
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001A0FR01
Record Dates: First submitted 2022-10-27; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Chronic Myeloid Leukemia
Keywords: BCR::ABL,; Chronic myeloid leukemia,; Tyrosine kinase inhibitor,; T315I mutation
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- 3L+ Cohort: Patients who initiated third-line treatment (3L) therapy. Treatments received in 3L were dasatinib, nilotinib, imatinib, ponatinib, bosutinib, and allo-SCT
  Interventions: Other: 3L Therapy
- T315I cohort: Patients with chronic myeloid leukemia with T315I mutation
  Interventions: Other: T315I

INTERVENTIONS:
Other: 3L Therapy — Treatments received in 3L were dasatinib, nilotinib, imatinib, ponatinib, bosutinib, and allo-SCT
  Other Names: third-line treatment
  Groups: 3L+ Cohort
Other: T315I — Patients with chronic myeloid leukemia with T315I mutation
  Groups: T315I cohort

SUMMARY:
A retrospective multi-center cohort study design was used to address the study objectives, using medical records obtained from three clinical centers in France.

DETAILED DESCRIPTION:
The index date for patients in the 3L cohort was defined as the date of initiation of 3L therapy. The index date for the T315I cohort was defined as the date of treatment initiation with TKI or allogeneic stem cell transplantation (allo-SCT) after identification of T315I mutation status. The baseline (i.e., pre-index) period was defined as the 6 months prior to the index date, and the post-index period was defined as the time from the index date to the date of last patient contact or patient death. Patients who were alive at the end of the follow-up period were censored at the date of last contact.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CML-CP
* Age ≥18 years at the time of CML-CP diagnosis
* For 3L patients: initiated one of the following 3L therapies in CML-CP after failing on ≥2 TKIs (i.e., bosutinib, dasatinib, imatinib, nilotinib, or ponatinib) or allo-SCT
* For T315I mutation patients: evidence of T315I mutation and treatment with TKI or allo-SCT

Exclusion Criteria:

* History of other active malignancies within the 3 years prior to the time of CML-CP diagnosis
* Documentation of anti-cancer therapies for any other malignancies prior to the time of 3L therapy initiation or at the time of treatment initiation after identification of T315I mutation
* Enrollment in a clinical trial at the time of 3L therapy initiation or at the time of treatment initiation after identification of T315I mutation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included CML-CP patients (i.e., 3L patients and patients with T315I mutation) who met the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Number of patients: Year patient initiated third-line treatment | throughout the study (study used data from 2000 to 2021)
  Following categories included:
  Before 2010 2010-2014 2015-2019 2020-2021
Duration of third-line treatment | throughout the study (study used data from 2000 to 2021)
  Duration of third-line treatment was reported
Number of patients: Type of therapy received in third-line treatment | throughout the study (study used data from 2000 to 2021)
  * TKI agent
  * Allo-SCT
Time from 2L discontinuation to third-line treatment initiation | throughout the study (study used data from 2000 to 2021)
  Time from 2L discontinuation to third-line treatment initiation was reported
Number of patients still on 3L therapy as of data collection date | throughout the study (study used data from 2000 to 2021)
  Number of patients still on 3L therapy as of data collection date was reported
Number of patients discontinued 3L | throughout the study (study used data from 2000 to 2021)
  Number of patients who discontinued 3L treatment were reported
Number of patients: Reasons for 3L discontinuation | throughout the study (study used data from 2000 to 2021)
  * Treatment switch due to AEs or intolerance
  * Treatment switch due to resistance
  * Treatment switch due to signs of ineffectiveness
  * Treatment switch due to other reasons
Number of lines of therapy for patients with chronic myeloid leukemia in third-line treatment | throughout the study (study used data from 2000 to 2021)
  Number of lines of therapy for patients with chronic myeloid leukemia in third-line treatment were reported
Number of most frequent treatment sequences for patients with chronic myeloid leukemia in third-line treatment | throughout the study (study used data from 2000 to 2021)
  Number of most frequent treatment sequences for patients with chronic myeloid leukemia in third-line treatment were reported
Number of last line of therapy for patients with chronic myeloid leukemia in third-line treatment | throughout the study (study used data from 2000 to 2021)
  Number of last line of therapy for patients with chronic myeloid leukemia in third-line treatment were reported
Number of patients: Year patient initiated on the line identified as T315I line of interest | throughout the study (study used data from 2000 to 2021)
  Following categories included:
  Before 2010 2010-2014 2015-2019
Duration of the line identified as T315I line of interest | throughout the study (study used data from 2000 to 2021)
  Duration of the line identified as T315I line of interest was reported
Number of patients: Type of therapy received in the line identified as T315I line of interest | throughout the study (study used data from 2000 to 2021)
  * TKI agent
  * Allo-SCT
Number of patients still on line of therapy identified as T315I line of interest as of data collection date | throughout the study (study used data from 2000 to 2021)
  Number of patients still on line of therapy identified as T315I line of interest as of data collection date were reported
Number of patients: Reasons for discontinuation on the line identified as T315I line of interest | throughout the study (study used data from 2000 to 2021)
  * Adverse events or intolerance
  * Resistance
  * Signs of ineffectiveness Suboptimal response Progression to accelerated phase or blast phase
  * Other reasons Acquired mutations
Number of lines of therapy for patients with chronic myeloid leukemia with T315I mutation | throughout the study (study used data from 2000 to 2021)
  Number of lines of therapy for patients with chronic myeloid leukemia with T315I mutation were reported
Number of line identified as T315I line of interest | throughout the study (study used data from 2000 to 2021)
  Number of line identified as T315I line of interest were reported
Number of treatment sequence for patients with chronic myeloid leukemia with T315I mutation | throughout the study (study used data from 2000 to 2021)
  Number of treatment sequence for patients with chronic myeloid leukemia with T315I mutation were reported
Number of last line of therapy for patients with chronic myeloid leukemia with T315I mutation | throughout the study (study used data from 2000 to 2021)
  Number of last line of therapy for patients with chronic myeloid leukemia with T315I mutation were reported

SECONDARY OUTCOMES:
Cytogenetic response (CyR) for 3L patients | 12 and 24 months
  CCyR, defined as an absence of Philadelphia chromosome-positive (Ph+) metaphases in bone marrow cytogenetics
Proportion of patients achieving response among patients with chronic myeloid leukemia in third-line treatment in 12 months | 12 months post treatment
  Proportion of patients achieving response among patients with chronic myeloid leukemia in third-line treatment in 12 months were reported
Proportion of patients achieving response among patients with chronic myeloid leukemia in third-line treatment in 24 months | 24 months post treatment
  Proportion of patients achieving response among patients with chronic myeloid leukemia in third-line treatment in 24 months were reported.
Proportion of patients achieving sustained molecular responses among patients with chronic myeloid leukemia in third-line treatment in 12 months | 12 months post treatment
  Proportion of patients achieving sustained molecular responses among patients with chronic myeloid leukemia in third-line treatment in 12 months were reported.
Proportion of patients achieving sustained molecular responses among patients with chronic myeloid leukemia in third-line treatment in 24 months | 24 months post treatment
  Proportion of patients achieving sustained molecular responses among patients with chronic myeloid leukemia in third-line treatment in 24 months were reported.
Time to major molecular response (MMR) among patients with chronic myeloid leukemia in third-line treatment | 12, 24, 36, 48, 60, 72 and 84 months post treatment
  Time to MMR was defined as the time from third-line (3L) treatment initiation to the time patients achieved MMR (i.e., 0.01% IS < BCR::ABL1 transcript level ≤ 0.1% IS). Patients were censored at the earliest of treatment discontinuation or switch, loss to follow-up, end of data availability, or death.
Time to deep molecular response (MR4.0) among patients with chronic myeloid leukemia in third-line treatment | 12, 24, 36, 48, 60, 72 and 84 months post treatment
  Time to MR4.0 was defined as the time from third-line (3L) treatment initiation to the time patients achieved MR4.0 (i.e., 0.0032% IS < BCR::ABL1 transcript level ≤ 0.01% IS). Patients were censored at the earliest of treatment discontinuation or switch, loss to follow-up, end of data availability, or death.
Time to sustained deep molecular response (MR4.0) among patients with chronic myeloid leukemia in third-line treatment | 12, 24, 36, 48, 60, 72 and 84 months post treatment
  Time to sustained MR4.0 was defined as the time from third-line (3L) treatment initiation to the time patients achieved sustained MR4.0 or better (i.e., BCR::ABL1 ≤ 0.01%) in all consecutive assessments performed for at least 12 months (i.e., 365.25 days). Patients were censored at the earliest of treatment discontinuation or switch, loss to follow-up, end of data availability, or death.
Time to deep molecular response (MR4.5) among patients with chronic myeloid leukemia in third-line treatment | 12, 24, 36, 48, 60, 72 and 84 months post treatment
  Time to MR4.5 was defined as the time from third-line (3L) treatment initiation to the time patients achieved MR4.5 (i.e., 0.001% IS ≤ BCR::ABL1 transcript level ≤ 0.0032% IS). Patients were censored at the earliest of treatment discontinuation or switch, loss to follow-up, end of data availability, or death.
Time to sustained deep molecular response (MR4.5) among patients with chronic myeloid leukemia in third-line treatment | 12, 24, 36, 48, 60, 72 and 84 months post treatment
  Time to sustained MR4.5 was defined as the time from third-line (3L) treatment initiation to the time patients achieved sustained MR4.5 or better (i.e., BCR::ABL1 ≤ 0.0032%) in all consecutive assessments performed for at least 2 years (i.e., 730.5 days). Patients were censored at the earliest of treatment discontinuation or switch, loss to follow-up, end of data availability, or death.
Time to Progression-free survival (PFS) for 3L patients | 12, 24, 36, 48, 60, 72 and 84 months post treatment
  Time to PFS was defined as the time from third-line treatment initiation to earliest occurrence of documented disease progression to accelerated phase or blast crisis, or the date of death from any cause. Patients were censored at the earliest of treatment discontinuation or switch, loss to follow-up, or end of data availability.
Time to Overall Survival (OS) for 3L patients | 12, 24, 36, 48, 60, 72 and 84 months post treatment
  Time to OS was defined as the time from third-line treatment initiation to death from any cause. Patients were censored at the earliest of treatment discontinuation or switch, date of last follow-up, or end of data availability.
Time to treatment discontinuation (TTD) for 3L patients | 12, 24, 36, 48, 60, 72 and 84 months post treatment
  TTD was defined as the time from third-line treatment initiation to treatment discontinuation or switch. Patients were censored at the earliest of loss to follow-up, or end of data availability, or death
Proportion of patients with Adverse Events (AEs) in third-line treatment | throughout the study (study used data from 2000 to 2021)
  Proportion of patients with Adverse Events (AEs) were reported to evaluate the safety profile of third-line treatments for chronic myeloid leukemia
Age of patients with chronic myeloid leukemia in third-line treatment | Index date defined as the date of initiation of 3L therapy (data from 2000 to 2021)
  Age information was reported.
Number of patients: Year of chronic myeloid leukemia in chronic phase (CML-CP) diagnosis of patients with chronic myeloid leukemia in third-line treatment | throughout the study (study used data from 2000 to 2021)
  Year of CML-CP diagnosis of patients with chronic myeloid leukemia in third-line treatment was reported.
Sex of patients with chronic myeloid leukemia in third-line treatment | Index date defined as the date of initiation of 3L therapy (data from 2000 to 2021)
  Sex information was reported.
Number of patients: Medical center of patients with chronic myeloid leukemia in third-line treatment | Index date defined as the date of initiation of 3L therapy (data from 2000 to 2021)
  The following centers were included:
  Centre Léon Bérard, Lyon Hématologie Institut Bergonié, Bordeaux Institut Universitaire du Cancer Toulouse, Toulouse
Length of follow-up (month) characteristics of patients with chronic myeloid leukemia in third-line treatment | throughout the study (study used data from 2000 to 2021)
  Length of follow-up was defined as time from index date to the date of last known contact with patient or patient death.
Number of patients: Smoking status at index date of patients with chronic myeloid leukemia in third-line treatment | Index date defined as the date of initiation of 3L therapy (data from 2000 to 2021)
  Smoking status at index date of patients with chronic myeloid leukemia in third-line treatment was reported.
Time from CML-CP diagnosis to index date (month) of patients with chronic myeloid leukemia in third-line treatment | throughout the study (study used data from 2000 to 2021)
  Time from CML-CP diagnosis to index date (month) of patients with chronic myeloid leukemia in third-line treatment was reported.
Number of patients with Hasford score at CML-CP diagnosis (month) of patients with chronic myeloid leukemia in third-line treatment | throughout the study (study used data from 2000 to 2021)
  Low risk (≤780) Intermediate risk (>780 to ≤1480) High risk (>1480) Not assessed Unknown / not sure
Number of patients with Sokal score at CML-CP diagnosis (month) of patients with chronic myeloid leukemia in third-line treatment | throughout the study (data source from 2000 to 2021)
  Low risk (<0.8) Intermediate risk (≥0.8 to ≤1.2) High risk (>1.2) Not assessed Unknown / not sure
Number of patients with ELTS risk score at CML-CP diagnosis (month) of patients with chronic myeloid leukemia in third-line treatment | throughout the study (data source from 2000 to 2021)
  ELTS: EUTOS long-term survival Low risk (≤1.5680) Intermediate risk (>1.5680 to ≤2.2185) High risk (>2.2185) Not assessed Unknown / not sure
Number of patients with BCR::ABL1 rearrangement at CML-CP diagnosis of patients with chronic myeloid leukemia in third-line treatment | throughout the study (data source from 2000 to 2021)
  Major Minor Other
Number of patients with Additional chromosomal abnormalities at CML-CP diagnosis of patients with chronic myeloid leukemia in third-line treatment | throughout the study (study used data from 2000 to 2021)
  Yes No
Number of comorbid conditions prior to the index date in patients with chronic myeloid leukemia in third-line treatment | Baseline (6 months prior to index date, defined as the date of initiation of 3L therapy)
  Number of comorbid conditions prior to the index date in patients with chronic myeloid leukemia in third-line treatment were reported.
Number of patients with comorbid conditions prior to the index date in patients with chronic myeloid leukemia in third-line treatment | Baseline (6 months prior to index date, defined as the date of initiation of 3L therapy)
  Cardiovascular disease Pulmonary disease/pulmonary arterial hypertension Gastrointestinal issues Renal disease Diabetes Liver disease Other No comorbidities Unknown / not sure
Number of patients with any ischemic condition prior to the index date in patients with chronic myeloid leukemia in third-line treatment | Baseline (6 months prior to index date, defined as the date of initiation of 3L therapy)
  Cardiovascular disease Cerebrovascular disease Peripheral arterial
Number of patients with Cardiovascular risk factors prior to the index date in patients with chronic myeloid leukemia in third-line treatment | Baseline (6 months prior to index date, defined as the date of initiation of 3L therapy)
  Hypertension Hyperlipidemia/dyslipidemia Diabetes Obesity
Laboratory and clinical results: Random blood glucose (mg/dl) | throughout the study (study used data from 2000 to 2021)
  Laboratory and clinical results were reported.
Laboratory and clinical results: Fasting blood glucose (mg/dl) | throughout the study (study used data from 2000 to 2021)
  Laboratory and clinical results were reported.
Laboratory and clinical results: LDL cholesterol (mg/dl) | throughout the study (study used data from 2000 to 2021)
  Laboratory and clinical results were reported.
Laboratory and clinical results: Total cholesterol (mg/dl) | throughout the study (study used data from 2000 to 2021)
  Laboratory and clinical results were reported.
Laboratory and clinical results: Blood pressure | throughout the study (study used data from 2000 to 2021)
  Laboratory and clinical results were reported.
Laboratory and clinical results: Spleen size below costal margin | throughout the study (study used data from 2000 to 2021)
  Laboratory and clinical results were reported.
Laboratory and clinical results: Blood cell count | throughout the study (study used data from 2000 to 2021)
  Laboratory and clinical results were reported.
Laboratory and clinical results: Bone marrow differential cell count | throughout the study (study used data from 2000 to 2021)
  Laboratory and clinical results were reported.
Number of patients with BCR::ABL1 mutation status by line of therapy for patients with chronic myeloid leukemia in third-line treatment | throughout the study (study used data from 2000 to 2021)
  Laboratory and clinical results were reported.
Proportion of patients achieving response among patients with chronic myeloid leukemia with T315I mutation | throughout the study (study used data from 2000 to 2021)
  Laboratory and clinical results were reported.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Lyon, France

IPD SHARING:
Plan to Share IPD: No